CLINICAL TRIAL: NCT01374906
Title: A Randomized, Double-blind, Multicenter, Phase III Study to Evaluate the Efficacy and Safety of Pasireotide LAR in Patients With Cushing's Disease
Brief Title: Efficacy and Safety of Pasireotide Administered Monthly in Patients With Cushing's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSOM230G2304; 2009-011128-70 (EudraCT Number)
Record Dates: First submitted 2011-06-14; First posted 2011-06-16 (Estimated); Results first posted 2018-04-11 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-04

CONDITIONS: Cushing's Disease
Keywords: SOM230; Cushing's Disease; Mean Urinary Free Cortisol; Pasireotide; Pasireotide LAR; Pasireotide long-acting release; secondary hypercortisolism; secondary hypercorticism; Itsenko-Cushing disease; increased secretion of adrenocorticotropic hormone (ACTH); hyperpituitarism
MeSH Terms: conditions — Pituitary ACTH Hypersecretion; Hyperpituitarism | interventions — pasireotide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 10 mg LAR dose (Experimental): Randomization was stratified based on Screening mUFC to ensure balanced distribution of disease severity in the two dose arms.
  Interventions: Drug: pasireotide LAR; Drug: SOM230 LAR 10 mg
- 30 mg LAR dose (Experimental): Randomization was stratified based on Screening mUFC to ensure balanced distribution of disease severity in the two dose arms.
  Interventions: Drug: pasireotide LAR; Drug: SOM230 LAR 30 mg

INTERVENTIONS:
Drug: pasireotide LAR — Pasireotide long-acting was administered as an intra-muscular depot intragluteal injection once every 28 days (±2 days). Patients were administered pasireotide long-acting 10 mg or 30 mg for four months, followed by either continuation of the starting dose, or dose up-titration (if mUFC was still >1.5xULN unless titration was precluded by safety reasons).
  Other Names: SOM230
Drug: SOM230 LAR 30 mg — starting dose of 30 mg i.m. administered once every 28 days for 4 months, followed by dose up-titration or continuation of starting dose.
  Arms: 30 mg LAR dose
Drug: SOM230 LAR 10 mg — starting does of SOM230 LAR 10 mg i.m. administered once every 28 days for 4 months, followed by dose up-titration or continuation of the starting dose.
  Arms: 10 mg LAR dose

SUMMARY:
This is a randomized, double-blind, multicenter, phase III study to evaluate the safety and efficacy of 2 dosing regiments of Pasireotide long acting release (LAR) in patients with Cushing's disease.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky performance status ≥ 60 (i.e. requires occasional assistance, but is able to care for most of their personal needs)
* For patients on medical treatment for Cushing's disease the following washout periods must be completed before screening assessments are performed

  * Inhibitors of steroidogenesis (ketoconazole, metyrapone): 1 week
  * Pituitary directed agents: Dopamine agonists (bromocriptine, cabergoline) and PPARγ agonists (rosiglitazone or pioglitazone): 4 weeks
  * Octreotide LAR, Lanreotide SR and Lanreotide autogel: 14 weeks
  * Octreotide (immediate release formulation): 1 week

Exclusion Criteria:

* Patients who are considered candidates for surgical treatment at the time of study entry
* Patients who have received pituitary irradiation within the last ten years prior to visit 1
* Patients who have had any previous pasireotide treatment
* Patients who have been treated with mitotane during the last 6 months prior to Visit 1
* Diabetic patients on antihyperglycemic medications with poor glycemic control as evidenced by HbA1c >8%
* Patients with risk factors for torsade de pointes, i.e. patients with a baseline QTcF >470 ms, hypokalemia, uncontrolled hypothyroidism, family history of long QT syndrome, or concomitant medications known to prolong QT interval
* Female patients who are pregnant or lactating, or are of childbearing potential (defined as all women physiologically capable of becoming pregnant) and not practicing an effective method of contraception/birth control. Sexually active males must use a condom during intercourse while taking the drug and for 2 months after the last dose of study drug and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-11-04 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (79):
- United States (12):
  - ClinTriCo, Phoenix, Arizona
  - University of California at Los Angeles UCLA Tiverton, Los Angeles, California
  - Harbor-UCLA Medical Center LA Biomed, Torrance, California
  - Emory University School of Medicine/Winship Cancer Institute G2304 - C2301, Atlanta, Georgia
  - Pituitary Center, Division of Endocrinology SC, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center SC-2, Ann Arbor, Michigan
  - Mount Sinai School of Medicine Mt. Sinai Medical Center, New York, New York
  - Oregon Health & Sciences University DeptofOregonHealth&Sciences(2), Portland, Oregon
  - University of Pennsylvania - Clinical Studies Unit Unniv SC, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center CSOM230G2304, Nashville, Tennessee
  - Swedish Medical Center Swedish, Seattle, Washington
  - Medical College of Wisconsin MCW 2, Milwaukee, Wisconsin
- Argentina (2):
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Córdoba
- Belgium (5):
  - Novartis Investigative Site, Edegem, Antwerpen
  - Novartis Investigative Site, Jette, Brussels Capital
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Brazil (4):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Ribeirão Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (3):
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Sherbrooke, Quebec
- China (3):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Shanghai
- France (6):
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Caen Cedex9
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille Cédex 5
  - Novartis Investigative Site, Pessac
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Germering
  - Novartis Investigative Site, Würzburg
- India (3):
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Vellore, Tamil Nadu
  - Novartis Investigative Site, New Delhi
- Novartis Investigative Site, Petah Tikva, Israel
- Italy (4):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Napoli
- Japan (12):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Nankoku, Kochi
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Osaka
- Novartis Investigative Site, Rotterdam, Netherlands
- Peru (2):
  - Novartis Investigative Site, Jesus Maria, Lima region
  - Novartis Investigative Site, Miraflores, Lima region
- Poland (4):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Spain (3):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Alzira, Valencia
  - Novartis Investigative Site, Barcelona
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Diskapi / Ankara, Ankara
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Izmir
- United Kingdom (4):
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Sheffield
  - Novartis Investigative Site, Southampton

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Lacroix A, Bronstein MD, Schopohl J, Delibasi T, Salvatori R, Li Y, Barkan A, Suzaki N, Tauchmanova L, Ortmann CE, Ravichandran S, Petersenn S, Pivonello R. Long-acting pasireotide improves clinical signs and quality of life in Cushing's disease: results from a phase III study. J Endocrinol Invest. 2020 Nov;43(11):1613-1622. doi: 10.1007/s40618-020-01246-0. Epub 2020 May 8. PMID 32385851
- [Derived] Newell-Price J, Pivonello R, Tabarin A, Fleseriu M, Witek P, Gadelha MR, Petersenn S, Tauchmanova L, Ravichandran S, Gupta P, Lacroix A, Biller BMK. Use of late-night salivary cortisol to monitor response to medical treatment in Cushing's disease. Eur J Endocrinol. 2020 Feb;182(2):207-217. doi: 10.1530/EJE-19-0695. PMID 31804965
- [Derived] Fleseriu M, Petersenn S, Biller BMK, Kadioglu P, De Block C, T'Sjoen G, Vantyghem MC, Tauchmanova L, Wojna J, Roughton M, Lacroix A, Newell-Price J. Long-term efficacy and safety of once-monthly pasireotide in Cushing's disease: A Phase III extension study. Clin Endocrinol (Oxf). 2019 Dec;91(6):776-785. doi: 10.1111/cen.14081. Epub 2019 Oct 1. PMID 31465533
- [Derived] Lacroix A, Gu F, Gallardo W, Pivonello R, Yu Y, Witek P, Boscaro M, Salvatori R, Yamada M, Tauchmanova L, Roughton M, Ravichandran S, Petersenn S, Biller BMK, Newell-Price J; Pasireotide G2304 Study Group. Efficacy and safety of once-monthly pasireotide in Cushing's disease: a 12 month clinical trial. Lancet Diabetes Endocrinol. 2018 Jan;6(1):17-26. doi: 10.1016/S2213-8587(17)30326-1. Epub 2017 Oct 12. PMID 29032078
- [Derived] Silverstein JM. Hyperglycemia induced by pasireotide in patients with Cushing's disease or acromegaly. Pituitary. 2016 Oct;19(5):536-43. doi: 10.1007/s11102-016-0734-1. PMID 27405306

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At least 148 patients (Pts.) were planned & 150 were randomized & analyzed. Pts. were all treated with either pasireotide long-acting 10 mg or pasireotide long-acting 30 mg. 81 Pts. completed the Core phase & entered the Extension phase with 39 completing the Extension phase.
Groups:
- 10 mg Pasireotide LAR Dose: Randomization was stratified based on Screening mUFC to ensure balanced distribution of disease severity in the two dose arms. These patients were dosed with 10 mg of Pasireotide LAR.
- 30 mg Pasireotide LAR Dose: Randomization was stratified based on Screening mUFC to ensure balanced distribution of disease severity in the two dose arms. These patients were dosed with 30 mg of Pasireotide LAR.
Period: Overall Study
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Started | 74 | 76
DC Dur Core Phs at/Prior to Data Cutoff | 24 | 22
Completed Core Phase | 50 | 54
Completed Core/Did Not Enter Ext. Phase | 10 | 13
Completed Core Phase/Entered Ext. Phase | 40 | 41
DC Dur Ext Phs at/Prior to Data Cutoff | 16 | 26
Completed Extension Phase | 24 | 15
Completed | 34 | 28
Not Completed | 40 | 48
Not completed — Abnormal laboratory value(s) | 0 | 3
Not completed — Administrative problems | 2 | 2
Not completed — Adverse Event | 10 | 11
Not completed — Death | 0 | 2
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 15 | 9
Not completed — Unsatisfactory therapeutic effect | 11 | 19

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose | Total
Number analyzed (Participants) | 74 | 76 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (12.52) | 38.6 (12.99) | 38.5 (12.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 60 | 118
  Male | 16 | 16 | 32
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 39 | 44 | 83
  Asian | 27 | 24 | 51
  Black | 2 | 0 | 2
  Other | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage Participants That Attained a mUFC ≤ 1.0 x ULN at Month 7 Regardless of Dose Titration
Description: Percentage of participants that attained a mean urinary free cortisol (mUFC) <= 1.0 x upper limit of normal (ULN) at Month 7 regardless of dose up-titration at Month 4. Patients who discontinued before month 4 evaluations classed as non-responders. For patients missing month 7 mUFC assessments, the last available mUFC assessment at or after month 4 was carried forward as the month 7 mUFC assessment value.
Time Frame: Month 7
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
percentage of participants | 41.9 [30.51 to 53.94] | 40.8 [29.65 to 52.67]

2. Secondary Outcome: Percentage of Participants That Attained a mUFC ≤ 1.0 x ULN at Month 7 and Had Not Had a Dose Increase at Month 4
Description: Percentage of participants that attain a mUFC ≤ 1.0×ULN at Month 7 and had not had a dose increase at Month 4. Patients who had a dose increase prior to Month 7 were counted as non-responders in this analysis.
  Patients who discontinued before month 4 evaluations classed as non-responders. For patients missing month 7 mUFC assessments, the last available mUFC assessment at or after month 4 was carried forward as the month 7 mUFC assessment value.
  A responder was defined as a patient who attains mUFC ≤1.0 X ULN and had not had a dose increase at Month 4.
Time Frame: Month 7
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
percentage of participants | 28.4 [18.50 to 40.05] | 31.6 [21.39 to 43.25]

3. Secondary Outcome: Actual Change in Mean Urinary Free Cortisol (mUFC) From Baseline
Description: Actual change in mUFC (nmol/24h) from baseline by randomized groups.
Time Frame: baseline, Month 7 (M7), Month 12 (M12), Month 24 (M24) , Month 36 (M36)
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: nmol/24h
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
nmol/24h
  M7: number analyzed (Participants) | 57 | 67
  M7 | -192.4 (271.59) | -234.3 (362.86)
  M12: number analyzed (Participants) | 50 | 54
  M12 | -195.1 (282.46) | -247.6 (387.05)
  M24: number analyzed (Participants) | 33 | 25
  M24 | -236.2 (292.91) | -265.2 (313.47)
  M36: number analyzed (Participants) | 14 | 4
  M36 | -398.4 (136.09) | -164.6 (66.76)

4. Secondary Outcome: Percentage Change in Mean Urinary Free Cortisol (mUFC) From Baseline
Description: Percentage change in mUFC (nmol/24h) from baseline by randomized groups.
Time Frame: M7, M12, M24, M36
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
percentage change
  M7: number analyzed (Participants) | 57 | 67
  M7 | -29.3 (102.76) | -33.2 (61.37)
  M12: number analyzed (Participants) | 50 | 54
  M12 | -30.3 (79.73) | -31.1 (78.41)
  M24: number analyzed (Participants) | 33 | 25
  M24 | -50.9 (76.48) | -51.2 (35.41)
  M36: number analyzed (Participants) | 14 | 4
  M36 | -71.6 (20.44) | -48.8 (11.36)

5. Secondary Outcome: Percentage of Patients Who Attain mUFC ≤ 1.0 x ULN
Description: Controlled responder: mUFC ≤ 1.0×ULN by randomized groups.
Time Frame: M7, M12, M24, M36
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
percentage of participants
  M7 - Controlled responder | 39.2 [28.04 to 51.23] | 40.8 [29.65 to 52.67]
  M12 - Controlled responder | 35.1 [24.39 to 47.11] | 25.0 [15.77 to 36.26]
  M24 - Controlled responder: number analyzed (Participants) | 63 | 61
  M24 - Controlled responder | 39.7 [27.57 to 52.80] | 21.3 [11.86 to 33.68]
  M36 - Controlled responder: number analyzed (Participants) | 50 | 50
  M36 - Controlled responder | 22.0 [11.53 to 35.96] | 4.0 [0.49 to 13.71]

6. Secondary Outcome: Percentage of Patients Who Attain mUFC ≤1.0 x ULN or Have at Least 50 % Reduction From Baseline in mUFC
Description: Controlled responder: mUFC ≤ 1.0×ULN. Partially controlled responder: at least 50% reduction in mUFC from Baseline, and mUFC >1.0×ULN.
Time Frame: M7, M12, M24, M36
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
percentage of participants
  M7 | 44.6 [33.02 to 56.61] | 53.9 [42.13 to 65.45]
  M12 | 45.9 [34.29 to 57.93] | 42.1 [30.86 to 53.98]
  M24: number analyzed (Participants) | 63 | 61
  M24 | 46.0 [33.39 to 59.06] | 27.9 [17.15 to 40.83]
  M36: number analyzed (Participants) | 50 | 50
  M36 | 28.0 [16.23 to 42.49] | 6.0 [1.25 to 16.55]

7. Secondary Outcome: Percentage of Patients Who Are Controlled Responders (mUFC ≤ 1.0 xULN) on at Least 4 of the 7 mUFC Assessments by Month 7 & on at Least 7 of the 12 mUFC Assessments by Month 12.
Description: Percentage of patients with mUFC ≤ 1.0 x ULN at a minimum of 4 months up to and including Month 7, and at a minimum of 7 months up to and including Month 12 by randomized groups.
Time Frame: Month 7, Month 12
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
percentage of participants
  Month 7 | 25.7 [16.22 to 37.16] | 31.6 [21.39 to 43.25]
  Month 12 | 25.7 [16.22 to 37.16] | 25.0 [15.77 to 36.26]

8. Secondary Outcome: Percentage of Patients With Uncontrolled Response at Month 7 & Month 12 Within the Subset of Patients Who Had Uncontrolled Response at a) Months 1 and 2; b) Months 1, 2, and 3
Description: Percentage of patients with mUFC > 1.0 xULN at Month 7 and Month 12 within the subset of patients who were uncontrolled at a) Months 1 & 2, b) Months 1, 2, & 3 by randomized groups.
Time Frame: Month 7, Month12
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
percentage of participants
  Uncontrolled Resp @ M7: subset: M1 & 2: number analyzed (Participants) | 33 | 33
  Uncontrolled Resp @ M7: subset: M1 & 2 | 60.6 | 60.6
  Uncontrolled Resp @ M7: subset: M1,2 & 3: number analyzed (Participants) | 31 | 29
  Uncontrolled Resp @ M7: subset: M1,2 & 3 | 61.3 | 65.5
  Uncontrolled Resp @ M12: subset: M1 & 2: number analyzed (Participants) | 33 | 33
  Uncontrolled Resp @ M12: subset: M1 & 2 | 69.7 | 69.7
  Uncontrolled Resp @ M12: subset: M1, 2 & 3: number analyzed (Participants) | 31 | 29
  Uncontrolled Resp @ M12: subset: M1, 2 & 3 | 74.2 | 72.4

9. Secondary Outcome: Percent of Participants Attaining a mUFC ≤ 1.0 x ULN or at Least a 50% Reduction in mUFC From Baseline at Indicated Time Points
Description: Time to first achievement of attaining a mUFC ≤ 1.0 x ULN or at least a 50% reduction in mUFC from baseline by randomized groups.
Time Frame: Momth 7, Month 12
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
Percentage of participants
  Month 7 | 86.2 [76.1 to 93.5] | 83.4 [72.6 to 91.8]
  Month 12 | 90.1 [80.7 to 96.2] | 94.5 [81.0 to 99.4]

10. Secondary Outcome: Percent of Participants Attaining a Duration of Controlled or Partially Controlled Response at Indicated Time Points
Description: Duration of controlled or partially controlled response is defined as the period starting from the date of patient's first normalization (mUFC≤ 1.0 x ULN) or at least 50% reduction from baseline up to the date when the patient's mUFC >1.0 x ULN and the reduction from baseline falls to less than 50% for the first time.
Time Frame: Month 6, 12, 18
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
Percentage of participants
  Month 6 | 78.0 [66.5 to 87.7] | 72.9 [61.2 to 83.4]
  Month 12 | 84.0 [73.1 to 92.2] | 82.8 [71.5 to 91.5]
  Month 18 | 84.0 [73.1 to 92.2] | 87.1 [74.6 to 95.3]

11. Secondary Outcome: Percentage Change From Baseline on Plasma Adrenocorticotropic Hormone (ACTH) Over Time
Description: Percentage change in ACTH (pmol/L) from Baseline by randomized groups.
Time Frame: Months 7, 12, 24 & 36
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
Percentage change
  M7: number analyzed (Participants) | 54 | 62
  M7 | 2.7 (57.14) | -13.5 (46.75)
  M12: number analyzed (Participants) | 44 | 52
  M12 | -10.2 (57.57) | -14.5 (38.72)
  M24: number analyzed (Participants) | 31 | 23
  M24 | -12.1 (43.51) | 2.5 (68.69)
  M36: number analyzed (Participants) | 13 | 5
  M36 | -15.4 (36.90) | -0.6 (48.13)

12. Secondary Outcome: Percentage Change From Baseline on Serum Cortisol Over Time
Description: Percentage change in serum cortisol (nmol/L) from Baseline by randomized groups.
Time Frame: Months 7, 12, 24 & 36
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
Percentage change
  M7: number analyzed (Participants) | 55 | 66
  M7 | -8.2 (37.83) | -5.1 (40.20)
  M12: number analyzed (Participants) | 46 | 54
  M12 | -12.1 (29.69) | -0.4 (35.91)
  M24: number analyzed (Participants) | 32 | 25
  M24 | -15.6 (30.67) | -7.4 (38.37)
  M36: number analyzed (Participants) | 14 | 5
  M36 | 0.6 (55.67) | -23.2 (31.19)

13. Secondary Outcome: Actual Change From Baseline in Clinical Signs Over Time: Blood Pressure
Description: Change in blood pressure measurements from Baseline
Time Frame: Month 7
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
mmHg
  Supine systolic blood pressure (SBP): number analyzed (Participants) | 57 | 67
  Supine systolic blood pressure (SBP) | -6.8 (15.64) | -4.6 (14.51)
  Supine diastolic blood (DBP) pressure: number analyzed (Participants) | 57 | 67
  Supine diastolic blood (DBP) pressure | -4.8 (12.06) | -3.0 (12.12)

14. Secondary Outcome: Actual Change From Baseline in Clinical Signs Over Time: Body Mass Index (BMI)
Description: Change in BMI measurements from Baseline
Time Frame: Month 7
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
kg/m2 | -0.7 (1.60) | -1.8 (2.05)

15. Secondary Outcome: Actual Change From Baseline in Clinical Signs Over Time: Weight
Description: Change in weight measurements from Baseline
Time Frame: Month 7
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
kg | -1.8 (4.16) | -4.6 (5.08)

16. Secondary Outcome: Actual Change From Baseline in Clinical Signs Over Time: Body Composition: Region
Description: Change in body composition: region measurements from Baseline
Time Frame: Month 7
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: percentage fat
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
percentage fat | -1.0 (2.64) | -1.8 (3.97)

17. Secondary Outcome: Actual Change From Baseline in Clinical Signs Over Time: Waist Circumference
Description: Change in waist circumference measurements from Baseline
Time Frame: Month 7
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
cm | -1.6 (8.47) | -7.1 (11.78)

18. Secondary Outcome: Actual Change From Baseline in Clinical Signs Over Time: Cholesterol & Triglycerides
Description: Change in parameter measurements: cholesterol & triglycerides from Baseline
Time Frame: Month 7
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
mmol/L
  Total cholesterol: number analyzed (Participants) | 56 | 64
  Total cholesterol | -0.5 (1.07) | -0.4 (1.00)
  HDL cholesterol: number analyzed (Participants) | 55 | 64
  HDL cholesterol | -0.1 (0.28) | 0 (0.32)
  Triglycerides: number analyzed (Participants) | 56 | 64
  Triglycerides | 0 (0.53) | -0.2 (0.64)

19. Secondary Outcome: Percentage Change From Baseline in Clinical Signs Over Time
Description: Percentage change in parameter measurements: blood pressure, body mass index, waist circumference, fasting serum lipid profile, weight, bone density and body composition (examined by DXA scan) from Baseline
Time Frame: Month 7
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
Percentage change
  SBP: number analyzed (Participants) | 57 | 67
  SBP | -4.3 (11.46) | -3.0 (10.18)
  DBP: number analyzed (Participants) | 57 | 67
  DBP | -4.7 (14.19) | -2.6 (13.78)
  BMI: number analyzed (Participants) | 57 | 67
  BMI | -2.6 (5.26) | -6.1 (6.94)
  Weight: number analyzed (Participants) | 57 | 67
  Weight | -2.6 (5.26) | -6.1 (6.91)
  Waist circumference: number analyzed (Participants) | 53 | 63
  Waist circumference | -1.4 (8.60) | -6.6 (10.06)
  HDL: number analyzed (Participants) | 55 | 64
  HDL | -6.7 (15.18) | 0.3 (20.91)
  Total cholesterol: number analyzed (Participants) | 56 | 64
  Total cholesterol | -7.2 (16.86) | -6.6 (16.40)
  Triglycerides: number analyzed (Participants) | 56 | 64
  Triglycerides | 4.2 (39.54) | -0.9 (39.61)
  Body composition: number analyzed (Participants) | 41 | 48
  Body composition | -2.4 (6.68) | -3.6 (10.47)

20. Secondary Outcome: Percentage of Participants Having a Favorable Shift From Baseline in Clinical Signs
Description: This includes patients with improvements in symptoms from baseline. Clinical signs over time include: facial rubor, fat pads, hirsutism, striae, (via photographs by a second local physician who was blinded to the treatment dose and time point of the photograph) and muscle strength.
Time Frame: Month 7
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
Percentage of participants
  Facial rubor: number analyzed (Participants) | 52 | 56
  Facial rubor | 32.7 | 53.6
  Hirsutism (females only): number analyzed (Participants) | 42 | 76
  Hirsutism (females only) | 22.2 | 32.6
  Striae: number analyzed (Participants) | 52 | 55
  Striae | 23.1 | 23.6
  Bruising: number analyzed (Participants) | 52 | 56
  Bruising | 25.0 | 14.3
  Supraclavicular fat pad: number analyzed (Participants) | 52 | 56
  Supraclavicular fat pad | 40.4 | 28.6
  Dorsal fat pad: number analyzed (Participants) | 52 | 55
  Dorsal fat pad | 28.8 | 40.0
  Muscle strength: number analyzed (Participants) | 56 | 66
  Muscle strength | 8.9 | 4.5

21. Secondary Outcome: Percentage of Participants That Attained a Mean Urinary Free Cortisol (mUFC) <= 1.0 x Upper Limit of Normal (ULN) at Month 7 Regardless of Dose Up-titration at Month 4.
Description: All of the participants who discontinued prior to month 4 evaluations were classed as non-responders. For participants missing month 7 mUFC assessments, the last available mUFC assessment at or after month 4 was carried forward as the month 7 mUFC assessment value.
  Analysis split by screening strata of mUFC Stratum 1: mUFC 1.5x to < 2.0 x ULN Stratum 2: mUFC 2.0x to <= 5.0 x ULN
Time Frame: Month 7
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
percentage of participants
  stratum:1.5 x ULN to < 2.0 x ULN: number analyzed (Participants) | 25 | 25
  stratum:1.5 x ULN to < 2.0 x ULN | 52.0 [31.31 to 72.20] | 52.0 [31.31 to 72.20]
  stratum:2.0 x ULN to <= 5.0 x ULN: number analyzed (Participants) | 49 | 51
  stratum:2.0 x ULN to <= 5.0 x ULN | 36.7 [23.42 to 51.71] | 35.3 [22.43 to 49.93]

22. Secondary Outcome: Percentage of Patients That Attain a Reduction of at Least 50% in mUFC From Baseline
Description: All of the participants who discontinued prior to month 4 evaluations were classed as non-responders. For participants missing month 7 mUFC assessments, the last available mUFC assessment at or after month 4 was carried forward as the month 7 mUFC assessment value.
  Analysis split by screening strata of mUFC
  Stratum 1:
Time Frame: Months 7, 12, 24 & 36
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
percentage of participants
  M7 | 35.1 [24.39 to 47.11] | 43.4 [32.08 to 55.29]
  M12 | 35.1 [24.39 to 47.11] | 38.2 [27.25 to 50.02]
  M24: number analyzed (Participants) | 24 | 14
  M24 | 83.3 [62.62 to 95.26] | 57.1 [28.86 to 82.34]
  M36: number analyzed (Participants) | 8 | 3
  M36 | 100 [63.06 to 100.00] | 33.33 [0.84 to 90.57]

23. Secondary Outcome: Percent of Participants Attaining a Time to First Achievement of at Least a 50% Reduction in mUFC From Baseline at Indicated Time Points
Description: Time to first achievement of a 5by randomized groups.0% reduction in mUFC from baseline
Time Frame: every month in the core phase and every 3 months in the extension phase) up to and including the cut-off date for the Month 12 CSR (10-Nov-2015)
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
Percentage of participants
  M7 | 80.5 [69.7 to 89.3] | 73.4 [62.4 to 83.4]
  M12 | 84.4 [74.0 to 92.3] | 80.7 [69.4 to 89.8]

24. Secondary Outcome: Percent of Participants With a Duration of at Least 50% Reduction in mUFC From Baseline at Indicated Time Points
Description: Duration of 50% reduction from baseline is defined as the period starting from the date of patient's first 50% reduction from baseline
Time Frame: Months 6, 12 & 18
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
Percentage of participants
  M6 | 78.4 [66.6 to 88.3] | 77.8 [66.0 to 87.7]
  M12 | 84.9 [73.7 to 93.1] | 83.7 [72.6 to 92.1]
  M18 | 84.9 [73.7 to 93.1] | 83.7 [72.6 to 92.1]

25. Secondary Outcome: Pharmacokinetic (PK) Parameter: Ctrough
Description: Pasireotide trough levels (Ctrough) was 1 of the parameters used for PK assessments. Ctrough is the pre-dose PK concentration with an elapsed time from previous injection of 28+/-2 days. All patients randomized to the study had at least 1 PK observation & were therefore included in the pharmacokinetic analysis set. PK observations with missing concentrations, missing dose, missing elapsed time or an elapsed time from previous injection outside of 28 ±2 days window were excluded. Given that SOM230 LAR was administered once a month, Ctrough was collected every 28 days and thus this provides a summary of Ctrough values provided by incident dose (last dose administered prior to PK sample collection), not by randomized dose, hence each column is equivalent to an incident dose & not an arm/group. Patients randomized to either 10mg or 30mg could be titrated down to 5mg due to safety, or titrated up to 40mg, hence the 4 incident doses/columns that were allowed per protocol during this study.
Time Frame: Days 29, 57, 85, 113, 141, 169, 197, 225, 253, 281, 309, 337
Population: Pharmacokinetic analysis set (PAS): The PAS consists of all randomized patients who have received at least one dose of study drug and had at least one post dosing PK assessment.
  Patients were analyzed according to incident dose (defined as the last dose prior to the PK sample).
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 5 mg Pasireotide LAR Dose: These patients were dosed with 5 mg of Pasireotide LAR to assess Pharmacokinetics (PK).
- 40 mg Pasireotide LAR Dose: These patients were dosed with 40 mg of Pasireotide LAR to assess Pharmacokinetics (PK).
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose | 5 mg Pasireotide LAR Dose | 40 mg Pasireotide LAR Dose
Number analyzed (Participants) | 65 | 64 | 5 | 44
ng/mL
  Day 29: number analyzed (Participants) | 65 | 64 | 0 | 0
  Day 29 | 2.03 (1.25) | 7.63 (4.58) |  |
  Day 57: number analyzed (Participants) | 57 | 61 | 1 | 0
  Day 57 | 2.35 (1.15) | 7.82 (4.22) | 0.83 (NA) — N/A = not enough patients on this day to derive data |
  Day 85: number analyzed (Participants) | 59 | 51 | 2 | 0
  Day 85 | 2.39 (1.32) | 8.56 (4.26) | 1.03 (0.63) |
  Day 113: number analyzed (Participants) | 51 | 49 | 3 | 0
  Day 113 | 2.40 (1.11) | 8.31 (3.87) | 1.29 (0.24) |
  Day 141: number analyzed (Participants) | 25 | 50 | 2 | 20
  Day 141 | 2.47 (0.94) | 7.88 (4.00) | 1.04 (0.68) | 10.7 (4.91)
  Day 169: number analyzed (Participants) | 29 | 51 | 2 | 22
  Day 169 | 2.47 (0.95) | 8.46 (3.51) | 2.01 (0.22) | 12.0 (5.08)
  Day 197: number analyzed (Participants) | 35 | 44 | 2 | 21
  Day 197 | 2.88 (1.29) | 9.13 (4.25) | 0.72 (0.39) | 11.9 (5.87)
  Day 225: number analyzed (Participants) | 22 | 28 | 3 | 34
  Day 225 | 2.68 (0.98) | 8.57 (4.70) | 1.19 (0.43) | 11.3 (5.18)
  Day 253: number analyzed (Participants) | 17 | 27 | 5 | 33
  Day 253 | 2.87 (1.57) | 9.00 (4.93) | 1.77 (0.88) | 12.1 (5.21)
  Day 281: number analyzed (Participants) | 13 | 16 | 3 | 44
  Day 281 | 3.36 (1.48) | 8.18 (4.23) | 1.24 (0.52) | 11.4 (5.85)
  Day 309: number analyzed (Participants) | 23 | 19 | 1 | 43
  Day 309 | 2.50 (0.99) | 9.34 (5.61) | 0.66 (NA) — N/A = not enough patients on this day to derive data | 12.0 (4.58)
  Day 337: number analyzed (Participants) | 21 | 15 | 3 | 41
  Day 337 | 3.07 (1.62) | 8.90 (4.37) | 1.91 (1.79) | 12.6 (6.21)

26. Secondary Outcome: Pharmacokinetic (PK) Parameter: Cmax
Description: Pasireotide peak levels (Cmax) was one of the parameters used for PK assessments. Cmax is the post-dose PK concentration with an elapsed time from the previous injection of 21+/-2 days. All patients randomized to the study had at least one PK observation and were therefore included in the pharmacokinetic analysis set (PAS). Cmax PK observations ("Day 20" and "Day 104") with an elapsed time from the previous injection outside of 21+/-2 days window were excluded. Given that SOM230 LAR was administered once a month, the Cmax were collected every 28 days in this study, thus this provides a summary of Cmax values provided by incident dose (last dose administered prior to PK sample collection), not by randomized dose, hence each column is equivalent to an incident dose and not an arm/group. Patients randomized to either the 10mg or 30mg could be titrated down to 5mg due to safety, or titrated up to 40mg, hence the 4 incident doses/columns that were allowed per protocol during this study.
Time Frame: Days 22, 106, 190
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 5 mg Pasireptide LAR Dose: These patients were dosed with 5 mg of Pasireotide LAR to assess Pharmacokinetics (PK).
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose | 5 mg Pasireptide LAR Dose | 40 mg Pasireotide LAR Dose
Number analyzed (Participants) | 67 | 69 | 3 | 22
ng/mL
  Day 22 (M 0.75): number analyzed (Participants) | 67 | 69 | 0 | 0
  Day 22 (M 0.75) | 3.0 (1.50) | 8.2 (3.99) |  |
  Day 106 (M 3.75): number analyzed (Participants) | 54 | 51 | 3 | 0
  Day 106 (M 3.75) | 3.3 (1.92) | 9.4 (3.72) | 1.7 (0.42) |
  Day 190 (M6.75): number analyzed (Participants) | 32 | 40 | 2 | 22
  Day 190 (M6.75) | 4.0 (1.73) | 10.0 (3.91) | 1.4 (0.78) | 12.1 (5.21)

27. Secondary Outcome: Actual Change in Standardized Score of Cushing's Disease HRQoL (CushingQOL) Score From Baseline
Description: CushingQol is a disease-specific patient-reported outcome instrument. It is a single-domain 12 item Cushing's disease quality of life instrument. The Cushing's syndrome quality of life (CushingQoL) questionnaire is a single domain questionnaire which includes 12 self-report items scored using a five point Likert scale anchored at (1=always/very much and 5=never/not at all). The patient is asked to report what they think or feel about their Cushing's syndrome and how much the illness has interfered in usual activities over the past 4 weeks. The total score is standardized on a 0-100 scale with lower scores indicating a greater impact on quality of life.
Time Frame: Months 7, 12, 24 & 36
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
scores on a scale
  M7: number analyzed (Participants) | 56 | 64
  M7 | 5.7 (15.97) | 7.8 (11.63)
  M12: number analyzed (Participants) | 47 | 53
  M12 | 6.4 (17.56) | 6.8 (14.42)
  M24: number analyzed (Participants) | 32 | 25
  M24 | 5.9 (15.56) | 8.7 (12.80)
  M36: number analyzed (Participants) | 13 | 4
  M36 | 1.4 (9.10) | 14.6 (5.10)

28. Secondary Outcome: Actual Change in SF-12v2 Score From Baseline - Mental Component Summary
Description: SF-12v2 General Health Survey is a general patient reported outcome instrument over time. It is scored to provide eight health domain scores (Bodily Pain (BP), General Health (GH), Physical Functioning (PF), Role-Physical (RP), Social Functioning (SF), Role-Emotional (RE), Vitality (VT) and Mental Health (MH)). These eight domain scores can be combined to form two summary scores reflecting overall physical and mental health: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). The analyses reported here focus on PCS and MCS scores. The domain scores use a norm-based score, which standardizes the scores with respect to the mean and standard deviation of a nationally representative sample of United States (US) adults. These are the scores on the original scale which have not been transformed in any way. The possible range of scores is 0 to 100, with higher scores representing better outcomes.
Time Frame: Months 7, 12 & 24
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
scores on a scale
  M7: number analyzed (Participants) | 33 | 37
  M7 | 4.1 (8.81) | 4.3 (8.05)
  M12: number analyzed (Participants) | 28 | 33
  M12 | 2.3 (9.97) | 3.3 (8.26)
  M24: number analyzed (Participants) | 9 | 5
  M24 | 3.3 (10.43) | 6.4 (2.53)

29. Secondary Outcome: Actual Change in SF-12v2 Score From Baseline - Physical Component Summary
Description: as for outcome 28
Time Frame: Months 7, 12 & 24
Population: Full analysis set (FAS): The FAS comprises all randomized patients who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose
Number analyzed (Participants) | 74 | 76
scores on a scale
  M7: number analyzed (Participants) | 33 | 37
  M7 | 1.9 (8.50) | -0.8 (7.46)
  M12: number analyzed (Participants) | 28 | 33
  M12 | 4.9 (5.56) | -0.5 (6.73)
  M24: number analyzed (Participants) | 9 | 5
  M24 | 5.3 (4.32) | -1.1 (5.54)

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse Events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit up to approximately 5 years.
Groups:
- All Patients: All Patients from both the 10 mg and 30 mg groups.
Arm/Group | 10 mg Pasireotide LAR Dose | 30 mg Pasireotide LAR Dose | All Patients
Serious Adverse Events (participants affected / at risk) | 22/74 | 19/76 | 41/150
Other Adverse Events (participants affected / at risk) | 73/74 | 76/76 | 149/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg Pasireotide LAR Dose (N=74) | 30 mg Pasireotide LAR Dose (N=76) | All Patients (N=150)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 1
Hyperadrenocorticism (Endocrine disorders) | 1 | 0 | 1
Pituitary-dependent Cushing's syndrome (Endocrine disorders) | 2 | 1 | 3
Anogenital dysplasia (Gastrointestinal disorders) | 1 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 1
Oedematous pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1
Injection site pain (General disorders) | 1 | 0 | 1
Malaise (General disorders) | 0 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 2 | 3 | 5
Cellulitis (Infections and infestations) | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 1 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 1
Stress fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2
Blood cortisol decreased (Investigations) | 1 | 1 | 2
Blood cortisol increased (Investigations) | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg Pasireotide LAR Dose (N=74) | 30 mg Pasireotide LAR Dose (N=76) | All Patients (N=150)
Anaemia (Blood and lymphatic system disorders) | 4 | 5 | 9
Palpitations (Cardiac disorders) | 4 | 3 | 7
Sinus bradycardia (Cardiac disorders) | 4 | 5 | 9
Vertigo (Ear and labyrinth disorders) | 5 | 0 | 5
Adrenal insufficiency (Endocrine disorders) | 4 | 6 | 10
Hypothyroidism (Endocrine disorders) | 1 | 4 | 5
Abdominal discomfort (Gastrointestinal disorders) | 4 | 2 | 6
Abdominal distension (Gastrointestinal disorders) | 4 | 5 | 9
Abdominal pain (Gastrointestinal disorders) | 11 | 13 | 24
Abdominal pain upper (Gastrointestinal disorders) | 3 | 8 | 11
Constipation (Gastrointestinal disorders) | 5 | 5 | 10
Diarrhoea (Gastrointestinal disorders) | 26 | 35 | 61
Dry mouth (Gastrointestinal disorders) | 4 | 1 | 5
Flatulence (Gastrointestinal disorders) | 3 | 5 | 8
Frequent bowel movements (Gastrointestinal disorders) | 4 | 0 | 4
Nausea (Gastrointestinal disorders) | 17 | 16 | 33
Vomiting (Gastrointestinal disorders) | 7 | 2 | 9
Asthenia (General disorders) | 10 | 5 | 15
Fatigue (General disorders) | 13 | 15 | 28
Oedema peripheral (General disorders) | 9 | 12 | 21
Pyrexia (General disorders) | 5 | 2 | 7
Cholelithiasis (Hepatobiliary disorders) | 15 | 33 | 48
Cholestasis (Hepatobiliary disorders) | 4 | 2 | 6
Gallbladder cholesterolosis (Hepatobiliary disorders) | 2 | 4 | 6
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 4 | 6
Hepatic steatosis (Hepatobiliary disorders) | 1 | 6 | 7
Bronchitis (Infections and infestations) | 5 | 2 | 7
Gastroenteritis (Infections and infestations) | 7 | 2 | 9
Influenza (Infections and infestations) | 12 | 6 | 18
Nasopharyngitis (Infections and infestations) | 18 | 13 | 31
Upper respiratory tract infection (Infections and infestations) | 5 | 6 | 11
Urinary tract infection (Infections and infestations) | 10 | 9 | 19
Contusion (Injury, poisoning and procedural complications) | 4 | 1 | 5
Alanine aminotransferase increased (Investigations) | 6 | 5 | 11
Blood cortisol decreased (Investigations) | 4 | 2 | 6
Blood creatine phosphokinase increased (Investigations) | 1 | 6 | 7
Blood glucose increased (Investigations) | 6 | 7 | 13
Gamma-glutamyltransferase increased (Investigations) | 7 | 6 | 13
Glycosylated haemoglobin increased (Investigations) | 4 | 4 | 8
Lipase increased (Investigations) | 2 | 4 | 6
Weight decreased (Investigations) | 4 | 3 | 7
Decreased appetite (Metabolism and nutrition disorders) | 3 | 12 | 15
Diabetes mellitus (Metabolism and nutrition disorders) | 15 | 20 | 35
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 6 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 36 | 35 | 71
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 4 | 5
Hyperuricaemia (Metabolism and nutrition disorders) | 5 | 5 | 10
Hypoglycaemia (Metabolism and nutrition disorders) | 10 | 12 | 22
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 4 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 4 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 8 | 16
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 5 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 6 | 12
Dizziness (Nervous system disorders) | 10 | 8 | 18
Headache (Nervous system disorders) | 18 | 10 | 28
Paraesthesia (Nervous system disorders) | 1 | 4 | 5
Insomnia (Psychiatric disorders) | 8 | 5 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 6
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 5 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 5 | 7
Erythema (Skin and subcutaneous tissue disorders) | 2 | 4 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 6 | 11
Rash (Skin and subcutaneous tissue disorders) | 4 | 2 | 6
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3 | 4 | 7
Hypertension (Vascular disorders) | 11 | 13 | 24
Hypotension (Vascular disorders) | 4 | 5 | 9

LIMITATIONS AND CAVEATS:
All analyses in this study were descriptive in nature. No comparisons were made between the two arms, and no p-values are reported. For the primary and key-secondary, success was based on estimating the response rate (and 95% CI) in each arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.